CLINICAL TRIAL: NCT05890677
Title: The LYMPH Trial - Comparing Microsurgical With Conservative Treatment of Chronic Breast Cancer Associated Lymphedema: Study Protocol of a Pragmatic Randomized International Multicentre Superiority Trial
Brief Title: The LYMPH Trial - Microsurgical Versus Conservative Treatment of Chronic Breast Cancer Associated Lymphedema
Acronym: LYMPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Rising Tide Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00733; mu21kappos; NCT07045831 (obsolete NCT alias)
Record Dates: First submitted 2023-05-23; First posted 2023-06-06 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Lymphedema, Breast Cancer
Keywords: lymphatic surgery; breast cancer related lymphedema; sentinel lymph node biopsy; axillary lymph node dissection; manual lymphatic drainage; conservative complex physical decongestion therapy
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Pragmatic, randomized, international, multicenter superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : Surgical Group (Experimental): According to the pragmatic study design, neither the diagnostic workup nor the surgery will be standardized in order to offer surgeons considerable leeway on how to perform lymphatic surgery, which resembles the flexibility in usual care. The key aspects of the preoperative workup and the surgery including the number of LVAs (Lymphovenous Anastomosis), harvesting of lymph nodes ("donor site"), time of surgery, and practical details will be registered.
  Interventions: Procedure: Surgical Intervention
- Group B: Conservative Complex Physical Decongestion Therapy (control group) (Active Comparator): CDT (Conservative Complex Physical Decongestion Therapy) will be performed as in usual care, following the pragmatic study design. The key aspects like frequency of lymphatic drainage, time when lymphatic drainage is performed and time and class of compressive garments are used will be documented. CDT incorporates two stages of treatment. The first treatment phase (intensive phase) entails skincare, MLD (manual lymphatic drainage), exercises aimed at improvement of mobility/range of motion in the shoulder, elbow or wrist joints, and compression therapy through bandaging. Most patients undergo this phase shortly after the diagnosis of LE. CDT in the second phase (maintenance phase) aims to maintain the achieved limb volume/ circumference reduction through compression with therapeutic elastic compression garment for the arm. Skincare, mobility exercises and MLD is continued in this phase if needed
  Interventions: Procedure: Conservative Complex Physical Decongestion Therapy

INTERVENTIONS:
Procedure: Surgical Intervention — LVA (Lymphovenous Anastomosis) and VLNT (Vascularised Lymph Node Transfer) are two advanced microsurgical techniques that are increasingly implemented in clinical practice in specialized centers and that are already carried out after health insurance application according to local standard of care. They have been studied in their respective mode of action as well as in their effectiveness in treating chronic BCRL (Breast Cancer-Related Lymphedema) in a multitude of mostly observational and single center studies with highly encouraging results. Patients in the interventional arm A will receive surgery with one of the two approaches or a combination of both, in a one or two-stage method, at the discretion of the treating surgeon. Depending on local standards one or both of the above might be combined with liposuction to the affected arm in a one or two-stage approach as well.
  Arms: Group A : Surgical Group
Procedure: Conservative Complex Physical Decongestion Therapy — Patients randomized to the control arm will receive CDT (Conservative Complex Physical Decongestion Therapy), which currently is considered as the best available standard of care. For this, patients will be referred to one of the dedicated LE (physical/skin) therapy clinics, if not already treated by one, according to their place of residence for continuation of standard conservative therapy. Recommendations to the procedures and treatment frequency of the conservative therapy will be made, but CDT will be done at the discretion of the treating physiotherapist.
  Arms: Group B: Conservative Complex Physical Decongestion Therapy (control group)

SUMMARY:
The aim of this study is to test whether lymphatic surgery provides better QoL (assessed with the Lymph-ICF-UL, (Lymphedema Functioning Disability and health questionnaire for upper limb lymphedema)) 15 months after randomization (and therefore about one year after surgery) compared to conservative treatment only for patients with chronic lymphedema (LE)

DETAILED DESCRIPTION:
To date, conservative complex physical decongestion therapy (CDT) is the gold standard for BCRL (breast cancer related lymphedema) and includes manual lymphatic drainage, local compression with bandages and garments, physical exercises and meticulous skin care. It is, however, too often ineffective to prevent stage progression in curing BCRL and purely symptomatic. Lymphovenous anastomosis (LVA) and vascularized lymph node transfer (VLNT) are two surgical techniques that, in contrast to CDT, are able to actually address the underlying causes and eventually restore the lymphatic drainage. LVA achieves this by creating numerous bypasses between lymphatic vessels and venules allowing the drainage of excessive fluid within the subcutaneous tissues into the venous system, while VLNT usually brings functioning lymph nodes to an area devoid of lymph nodes or with dysfunctional lymph nodes, thus enabling the spontaneous development of new lymphatic pathways. Both techniques have shown very promising results with low complication rates and improved Quality of Life (QoL) for the patients. However, no multicentric randomized controlled trial (RCT) has yet prospectively evaluated the superiority of these surgical techniques over CDT alone, limiting patient's access to most effective treatment available. Requests for cost reimbursement must still be submitted to insurance companies in most countries and are often rejected, thus delaying surgical treatment and resulting in prolonged suffering of affected patients. This is untenable seeing as affected patients suffer from a heavy physical, psychological and financial burden. This pragmatic, randomized, multicenter trial aims to establish a solid scientific basis assessing the superiority of surgical treatment over CDT alone.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients ≥ 18 years of age.
* Former diagnosis of breast cancer.
* Clinical diagnosis of chronic Breast Cancer-Related Lymphedema (BCRL) (persisting for more than 3 months) classified as ≥ Stage 1, according to ISL.
* Minimum of 3 months Conservative Complex Physical Decongestion Therapy.
* Ability to complete the QoL questionnaires.
* Willingness to undergo surgery.

Exclusion Criteria:

* No indication for lymphatic surgery according to clinical judgment of the treating surgeon (individual reasons will be specifically documented).
* Primary congenital Lymphedema or non-BCRL.
* Previous surgical BCRL treatment on the side intended for intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2036-06 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life Questionnaire (Lymph-ICF-UL) | two time assessment at baseline and 15 month after randomization
  The LYMPH-ICF-UL-Questionnaire (Lymphedema Functioning Disability and health questionnaire for upper limb lymphedema) is a widely used, rigorously developed, and validated patient-reported outcome (PRO) instrument for chronic breast cancer-related lymphedema. It assesses the impairments in function, activity limitations and participation restrictions of patients with upper limb lymphedema (LE). Consisting of 29 items (questions) across five different domains, each item is scored on a VAS (visual analog scale) ranging from 0 to 10. The total score on the LYMPH-ICF is equal to the sum of the item scores divided by the total number of answered items. A higher score on the Lymph-ICF indicates a greater impact on the functioning in daily life related to upper limb LE. This questionnaire helps determine if lymphatic surgery improves quality of life and patient satisfaction compared to conservative therapy.

SECONDARY OUTCOMES:
Change in Quality of Life Questionnaire (Lymph-ICF-UL) | 13 time assessment up to 10 years after randomization
  The LYMPH-ICF-UL-Questionnaire (Lymphedema Functioning Disability and health questionnaire for upper limb lymphedema) is a widely used, rigorously developed, and validated patient-reported outcome (PRO) instrument for chronic breast cancer-related lymphedema. It assesses the impairments in function, activity limitations and participation restrictions of patients with upper limb lymphedema (LE). Consisting of 29 items (questions) across five different domains, each item is scored on a VAS (visual analog scale) ranging from 0 to 10. The total score on the LYMPH-ICF is equal to the sum of the item scores divided by the total number of answered items. A higher score on the Lymph-ICF indicates a greater impact on the functioning in daily life related to upper limb LE. This questionnaire helps determine if lymphatic surgery improves quality of life and patient satisfaction compared to conservative therapy.
Change in Quality of Life Questionnaire (LYMPH-Q) | 15 time assessment up to 10 years after randomization
  The Lymph-Q Upper Extremity Module is a new PROM (patient-reported outcome measure) developed to assess patient reported outcomes of BCRL in a concept-driven approach. The complete questionnaire contains 68 questions covering the patient-relevant topics Health-related quality of life (arm appearance, arm function, arm symptoms, psychological), experience of care (information), and treatment (arm sleeve).
  The questionnaire is used to determine whether lymphatic surgery provides better quality of life and patient satisfaction compared to conservative therapy.
Change in Quality of Life Questionnaire (EuroQol EQ-5D-5L) | 15 time assessment up to 10 years after randomization
  The 5-level EQ-5D version (EQ-5D-5L) consists of the EQ-5D descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions (5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems) resulting in a 1-digit number that expresses the level for that dimension. The digits for each dimension can be combined into a 5-digit number that describes the patient's health state.
  The questionnaire is used to determine whether lymphatic surgery provides better quality of life and patient satisfaction compared to conservative therapy.
Change in Pain score (visual analog scale) | 7 time assessment up to 2 years after randomization
  The pain score consists of a VAS (visual analog scale) ranging from 0 (i.e. no pain) to 10 (i.e. worst pain). The VAS was published by the Yale University.
  It is used to determine whether lymphatic surgery provides better quality of life and patient satisfaction compared to conservative therapy.
Assessment of (serious) adverse events | 7 time assessment up to 2 years after randomization
  Safety is assessed via a rigorous and detailed examination of (serious) adverse events.
Assessment of surgical complications | 7 time assessment up to 2 years after randomization
  For the surgery group only, safety is assessed via a rigorous and detailed examination of complications of surgery. Grading is according to the modified classification of Clavien-Dindo, categorizing them into five levels ranging from minor deviations to life-threatening events.
  The assessment will cover both surgical stages in case of two-staged lymphedema (LE) surgery.
Assessment of lymphangitic events (erysipelas) | 7 time assessment up to 2 years after randomization
  The frequency of lymphangitic events (erysipelas) is closely monitored. Lymphangitic events are defined as skin infections at the lymphedema site(s) which can be treated with oral or intravenous antibiotics. The type of antibiotic given, the application form, type of hospital stay and necessity of a surgery will be assessed.
Assessment of arm volume | 15 time assessment up to 10 years after randomization
  Arm volume is determined by measuring the circumference of each arm at 10 cm intervals from the wrist to the axilla. The volume of each arm segment is calculated using a truncated cone model, and percentage edema volume is derived from the volume difference between the affected and unaffected arms. Both relative (relative to the unaffected arm) and absolute (volume reduction of the affected arm at the next measurement) volume change are calculated, corrected for BMI and differences between dominant and non-dominant arms.
Assessment of the frequency of lymphatic drainage | 15 time assessment up to 10 years after randomization
  The frequency of lymphatic drainage before the start of the study and between the study's follow-up visits is assessed.
Assessment of the burden on patients | 9 time assessment up to 10 years after randomization
  To assess the burden on patients, information regarding the total number of operative procedures, length of hospital stays, number of outpatient visits, and absence from work within two years after randomization and during the extended follow-up is collected.
Assessment of the economics (for Switzerland) | 9 time assessment up to 10 years after randomization
  To perform an economic evaluation, information regarding the condition-related medical resource use, healthcare costs, indirect costs, productivity losses, and incremental cost-effectiveness (quality-adjusted life-years) is collected.
  The information is based on the responses to the EQ-5D-5L questionnaire, the questions asked under burden on patients, and on other medical resource information recorded in the trial primarily for clinical purposes, at the respective visits. In addition, direct extraction of breast cancer-related lymphedema-related in- and outpatient costs, and corresponding key resource use parameters, are collected from the hospital administration systems of the participating Swiss sites, once at the 2 year follow-up visit .

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kappos, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (35):
- United States (4):
  - Yale School of Medicine, New Haven, Connecticut
  - Harvard Medical School, Boston, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Mayo Clinic, Rochester, New York
- Krankenhaus Göttlicher Heiland GmbH, Vienna, Austria
- Belgium (2):
  - Brussels University Hospital, Brussels, Jette
  - University of Ghent, Ghent
- Hospital Erasto Gaertner, Paraná, Curitiba, Brazil
- Canada (2):
  - McGill University, Royal Victoria Hospital, Montreal
  - University of British Columbia, Gordon and Leslie Diamond Health Care Centre, Vancouver
- Germany (9):
  - BG Universitätsklinikum Bergmannsheil Bochum, Bochum
  - Sana Kliniken Düsseldorf, Düsseldorf
  - Uniklinikum Erlangen, Erlangen
  - KEM Evang. Kliniken Essen-Mitte, Essen
  - BG Klinik Frankfurt am Main, Frankfurt
  - Universitätsklinikum Freiburg, Klinik für Plastische und Handchirurgie, Freiburg im Breisgau
  - BG Klinik Ludwigshafen, Ludwigshafen am Rhein
  - Klinikum Nürnberg, Nuremberg
  - Caritas Krankenhaus St. Josef/ Uniklinik Regensburg, Regensburg
- Papageorgiou Hospital of Thessaloniki, Thessaloniki, Greece
- Rambam Health Clinic, ISR, Haifa, Israel
- Italy (2):
  - Policlinico Tor Vergata: Fondazione PTV, Rome
  - Policlinico Universitario Fondazione Agostino Gemelli, Rome
- Maastricht University Medical Center, Maastricht, Netherlands
- Institute of Oncology ''Prof. Dr. Ion Chiricuță'' of Cluj-Napoca, Cluj-Napoca, Romania
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
- Sweden (2):
  - Karolinska Institutet, K1 Molekylär medicin och kirurgi, Stockholm
  - Department of Plastic and Reconstructive Surgery Uppsala University Hospital, Uppsala
- Switzerland (6):
  - Kantonsspital Aarau, Aarau
  - University Hospital Basel, Basel
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Winterthur, Winterthur
  - Klinik für Plastische, Rekonstruktive, Aesthetische und Handchirurgie, Zurich
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Metadata describing the type, size and content of the datasets will be shared along with the study protocol and case report forms on public repositories following FAIR (Findability, Accessibility, Interoperability and Reuse) principles. The DKF of the University of Basel will act as an independent Data Access Committee, storing the data at time of publication on secure servers, maintained and backed-up by the IT-department of the University Hospital Basel. Researchers can request data reuse by submitting a project synopsis via dkf.unibas.ch/contact. Study results will be published in peer-reviewed journals following the Consolidated Standards of Reporting Trials (CONSORT) standards for randomized controlled trials (RCTs) and good publication practice, regardless of outcomes. Authorship for future publications will be based on contributions. An annual safety report is submitted to the local Ethics Committee by the Sponsor-Investigator according to national regulations.

REFERENCES:
- [Derived] Kappos EA, Haas Y, Schulz A, Peters F, Savanthrapadian S, Stoffel J, Katapodi MC, Mucklow R, Kaiser B, Haumer A, Etter S, Cattaneo M, Staub D, Ribi K, Shaw J, Handschin TM, Eisenhardt S, Visconti G, Franceschini G, Scardina L, Longo B, Vetter M, Zaman K, Plock JA, Scaglioni M, Gonzalez EG, Quildrian SD, Felmerer G, Mehrara BJ, Ayala JM, Pons G, Kalbermatten DF, Sacks JM, Halle M, Muntean MV, Taylor EM, Mani M, Jung FJ, di Summa PG, Demiri E, Dionyssiou D, Groth AK, Heine N, Vorstenborsch J, Isaac KV, Qiu SS, Engels PE, Serre A, Eberhardt AL, Ebner S, Schwenkglenks M, Stoel Y, Leo C, Horch RE, Blondeel P, Behr B, Kneser U, Prantl L, Boll DT, Granziera C, Hemkens L, Lindenblatt N, Haug M, Schaefer DJ, Hirche C, Pusic AL, Seidenstuecker K, Harder Y, Weber W. The LYMPH trial: comparing microsurgical with conservative treatment for chronic breast cancer-associated lymphoedema - study protocol of a pragmatic randomised international multicentre superiority trial. BMJ Open. 2025 Feb 17;15(2):e090662. doi: 10.1136/bmjopen-2024-090662. PMID 39961719